CLINICAL TRIAL: NCT00001367
Title: Diagnosis and Natural History Protocol for Patients With Different Neurological Conditions
Brief Title: Diagnosis and History Study of Patients With Different Neurological Conditions
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930202; 93-N-0202
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-07

CONDITIONS: Nervous System Disease; Healthy Volunteer
Keywords: Healthy Volunteer; Nervous System Disease; Natural History
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- family members: Family Members who are 2 years old or older of people with a neurological disorder
- healthy volunteers: healthy volunteers age 18 and older
- patients: subjects with neurological disorders who are 2 years old or older

SUMMARY:
This protocol is a screening and natural history protocol, which allows for evaluation of

patients and families where neurological conditions are present for enrollment into other

studies and will also be used to screen healthy volunteers to create a pool of potential future HV matches for HMCS protocols. Through diagnostic evaluations, data will be collected for research use in this study.

...

DETAILED DESCRIPTION:
This protocol is a screening and natural history protocol, which allows for evaluation of

patients and families where neurological conditions are present for enrollment into other

studies and will also be used to screen healthy volunteers to create a pool of potential future HV matches for HMCS protocols. Through diagnostic evaluations, data will be collected for research use in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with neurological disorders and subjects with a family history of neurological conditions OR
* Healthy volunteers: People age 18 or older who are generally in good health.

EXCLUSION CRITERIA:

* Patients <2 years old.
* Employees of HMCS in NINDS.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The following population groups may participate: - Subjects with neurological disorders who are 2 years old or older, - Family members who are 2 years old or older of people with a neurological disorder, - Healthy volunteers who are 18 years old or older.
Sampling Method: Non-Probability Sample
Enrollment: 3813 (Actual)
Dates: Start 1993-09-30 (Actual)

PRIMARY OUTCOMES:
to screen patients with neurological conditions and family members of patients with neurological conditions for enrollment in additional research protocols | ongoing
  The goal is to screen patients with neurological conditions and family members of patients with neurological conditions for enrollment in additional research protocols. No investigational treatments will be administered on this protocol and the NIH physicians will be playing a consultative role to the patient s primary physician.

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This protocol was written before creating sharing plans was required. We do share data with other protocols done by our group to avoid having to repeat procedures, but there is no official "research" done in this protocol, so it is unlikely that we will need to share any IPD elsewhere. If there is, we will consider it on a case-by-case basis.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1993-N-0202.html